CLINICAL TRIAL: NCT04613687
Title: Evaluation of the Efficacy and Safety of a New Compression System URGO BD001 in the Treatment of Venous or Mixed Predominantly Venous Leg Ulcers
Brief Title: Efficacy and Safety of a New Compression System URGO BD001 in the Treatment of VLU (FREEDOM)
Acronym: FREEDOM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Laboratoires URGO (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FI-19-09-BD001
Record Dates: First submitted 2020-10-20; First posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer | interventions — Compression Bandages

STUDY DESIGN:
Intervention Model Description: Prospective, multi centre, non-comparative study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- URGOBD001 (Experimental): Compression bandage
  Interventions: Device: Compression bandage

INTERVENTIONS:
Device: Compression bandage — Compression bandage URGO BD001 for the management of venous leg ulcers with ABPI (Ankle Brachial Pressure Index) ≥ 0.8, venous

SUMMARY:
The aim of this study is to evaluate the therapeutic efficacy and the safety of the new compression system URGO BD001 in the management of venous or mixed predominantly venous leg ulcers. The therapeutic efficacy will be the reduction in wound surface area during a six weeks study treatment period.

DETAILED DESCRIPTION:
The compression bandage URGO BD001 is indicated for the management of venous leg ulcers with ABPI (Ankle Brachial Pressure Index) ≥ 0.8, venous oedema and lymphedema justifying strong compression.

The pressure applied with the compression system URGO BD001 help to improve venous return and to reduce venous oedema. The expected clinical benefits from the compression system URGO BD001 in patient with a VLU are to increase healing rate and time to healing, and to improve patient quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patient affected by VLU or mixed ulcer of predominantly venous origin (ankle brachial pressure index (ABPI) ≥ 0.8 and ≤ 1.3),
* Wound in granulation phase (granulation tissue ≥50%),
* Wound at least 3 cm away from any edge of another wound,
* VLU between 2 and 20 cm2 in surface area,
* VLU duration between 1 to 24 months.

Exclusion Criteria:

* Patient under guardianship or protection of vulnerable adult,
* Patient with known allergy to any components of the tested compression system,
* Patient with a severe illness that might lead to premature discontinuation of the trial before the end of treatment period,
* Patient with progressive neoplastic lesions treated by radiotherapy, chemotherapy, hormone therapy or immune suppressor,
* Patient with non-controlled systemic infection by a suitable antibiotic therapy,
* Patient who had a deep vein thrombosis within 3 months prior to the inclusion,
* Patient with a lymphedema due to lymphatic obstruction,
* Diabetic patient with advanced diagnosed microangiopathy,
* Bedridden patient, or those spending less than one hour per day on their feet,
* Wound covered partially or totally with necrotic tissue,
* Clinically infected wound,
* Wound requiring surgical treatment or for which a surgery is scheduled during the study period,
* Cancerous lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2020-10-30 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Relative reduction in wound surface area (percent) | 6 weeks
  Evolution between D0 and the 6 weeks treatment period with the URGO BD001 compression system: Relative reduction in wound surface area (%) = [(SW6 - SD0)/SD0] × 100 SD0: Wound surface area at D0 SW6: Wound surface area at Week 6

SECONDARY OUTCOMES:
Complete ulcer closure: | 6 weeks or last assessment
  The percent (%) of patients with complete ulcer closure (100% re-epithelialization) after 6 weeks or at the latest treatment period
Venous oedema | 6 weeks or last assessment
  Oedema reduction from baseline (D0) and last assessment by measuring the limb circumference (in cm), using a tape:
  * Ankle circumference at the reference point B (smallest perimeter of the leg, 3 cm above medial malleolus,
  * Calf circumference at the reference point C (maximum perimeter of the calf).
Patient quality of Life (EuroQoL 5D-5L) | 6 weeks or last assessment
  EuroQoL 5D-5L between baseline and at last visit. The questionnaire essentially consists of a descriptive system including 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression, and a visual analogue scale (EQ VAS) from "the worst health you can imagine" (0) to "the best health you can imagine" (100).
Evolution of the periwound skin | 6 weeks or last assessment
  Evolution of the peri-wound skin at each visit according to the following parameters:
  * Healthy
  * Altered: Erythematous and/or squamous (irritated dermatitis/eczema), maceration, other
Safety analysis | 6 weeks or last assessment
  Nature and number of adverse event related to the use of the testing compression system (serious/ non-serious)

CONTACTS AND LOCATIONS:
Overall Officials: Senet Patricia, MD, Principal Investigator — Vascular dermatologist, APHP, Paris, France; Dissemond Joachim, MD, Principal Investigator — Clinic for dermatology, Essen- Germany